CLINICAL TRIAL: NCT01534390
Title: The Influence of In-line Microfilters on Systemic Inflammation in Adult Critically Ill Patients: A Prospective, Randomized, Controlled Trial
Brief Title: Influence of In-line Microfilters on Systemic Inflammation in Adult Critically Ill Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Salzburg (Other)
Responsible Party: Principal Investigator, Martin W Duenser, MD, DESA, EDIC, Dr., University of Salzburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 415-E/1442/7-2012
Record Dates: First submitted 2012-02-09; First posted 2012-02-16 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Systemic Inflammation
Keywords: microparticles; in-line microfilters; systemic inflammation; organ failure; critical illness; adult
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Use of in-line microfilters (Experimental)
  Interventions: Device: In-line microfilter (Supor IV Filter; Pall Corporation, Port Washington, New York)
- Standard therapy without the use of in-line microfilters (No Intervention)

INTERVENTIONS:
Device: In-line microfilter (Supor IV Filter; Pall Corporation, Port Washington, New York) — use of in-line microfilters with a pore size of 0,2 mcm and 1,2 mcm (only if parenteral nutrition is administered) at all intravenous accesses
  Arms: Use of in-line microfilters

SUMMARY:
Studies showed that infusion or injection of drugs and fluids results in introduction of microparticles into the bloodstream. These microparticles may cause organ damage and stimulate the immune system thus aggravating the underlying disease. Given that critically ill patients are characteristically suffering from a high disease severity and receive large amounts of fluids and drugs, they may be at particular risk of harm by these microparticles. In-line microfilters have been shown to clear microparticles from intravenous drugs and solutions. The investigators hypothesize that use of in-line microfilters reduce the days with the systemic inflammatory response syndrome in adult critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* critical illness
* expected length of stay in the intensive care unit > 24 hours
* central venous catheter in place or placed within the first 24 hours

Exclusion Criteria:

* age < 18 years
* pregnancy
* neutropenia or known immunesuppresion
* limited intensive care
* inclusion into another clinical trial
* refusal of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of days in the intensive care unit with the systemic inflammatory response syndrome | participants will be followed for the duration of ICU stay, an expected average of 5 days

SECONDARY OUTCOMES:
Incidence of the systemic inflammatory response syndrome during the intensive care unit stay | participants will be followed for the duration of ICU stay, an expected average of 5 days
Average number of days with the systemic inflammatory response syndrome during the intensive care unit stay | participants will be followed for the duration of ICU stay, an expected average of 5 days
Length of stay in the intensive care unit | participants will be followed for the duration of ICU stay, an expected average of 5 days
Duration of mechanical ventilation | participants will be followed for the duration of ICU stay, an expected average of 5 days
Incidence of acute lung injury and the acute respiratory distress syndrome | participants will be followed for the duration of ICU stay, an expected average of 5 days
Maximum C-reactive protein serum concentrations during the intensive care unit stay | participants will be followed for the duration of ICU stay, an expected average of 5 days
Maximum leukocyte count during the intensive care unit stay | participants will be followed for the duration of ICU stay, an expected average of 5 days
Incidence of nosocomial infections during the intensive care unit stay | participants will be followed for the duration of ICU stay, an expected average of 5 days
Incidence of nosocomial candida infections during the intensive care unit stay | participants will be followed for the duration of ICU stay, an expected average of 5 days
Incidence of venous thrombosis during the intensive care unit stay | participants will be followed for the duration of ICU stay, an expected average of 5 days
Cumulative insulin requirements during the intensive care unit stay | participants will be followed for the duration of ICU stay, an expected average of 5 days
Number of days with hypo- or hyperglycemic blood sugar levels | participants will be followed for the duration of ICU stay, an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin W Duenser, MD, DESA, EDIC, Study Chair — Department of Anesthesiology, perioperative and intensive care medicine, Salzburg General Hospital and Paracelsus Private Medical University
Locations (1):
- Department of Anesthesiology, perioperative and intensive care medicine, Salzburg General Hospital and Paracelsus Private Medical University, Salzburg, Salzburg, Austria

REFERENCES:
- [Derived] Gradwohl-Matis I, Brunauer A, Dankl D, Wirthel E, Meburger I, Bayer A, Mandl M, Dunser MW, Grander W. Influence of in-line microfilters on systemic inflammation in adult critically ill patients: a prospective, randomized, controlled open-label trial. Ann Intensive Care. 2015 Dec;5(1):36. doi: 10.1186/s13613-015-0080-x. Epub 2015 Nov 4. PMID 26538309